CLINICAL TRIAL: NCT04294667
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Dapirolizumab Pegol in Study Participants With Moderately to Severely Active Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Efficacy and Safety of Dapirolizumab Pegol in Study Participants With Moderately to Severely Active Systemic Lupus Erythematosus
Acronym: PHOENYCS GO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0043; 2019-003406-27 (EudraCT Number)
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Dapirolizumab pegol; SLE; DZP
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapirolizumab pegol (Experimental): Subjects will receive dapriolizumab pegol througout the Treatment Period.
  Interventions: Drug: DZP
- Placebo (Placebo Comparator): Subjects will receive placebo througout the Treatment Period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DZP — Subjects will receive dapirolizumab pegol at prespecified time-points.
  Other Names: CDP7657
  Arms: Dapirolizumab pegol
Other: Placebo — Subjects will receive placebo at prespecified time-points.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the ability of dapirolizumab pegol (DZP) as an add-on treatment to standard of care (SOC) medication to achieve clinically relevant long term improvement of moderate to severe disease activity.

ELIGIBILITY:
Inclusion Criteria:

* Rescreening will be allowed once during the study in case there is new evidence for an inclusion criterion that was not fulfilled at the first screening or in case a study participant no longer meets an exclusion criterion or screening period exceeded the maximum duration due to delays in screening processes
* Study participant must be ≥16 years of age, unless restricted by local regulation, at the time of signing the Informed Consent form (ICF)
* Study participants who have moderate to severe disease activity due to either persisting active SLE or due to an acute worsening of SLE in the scope of frequent flaring/relapsing-remitting systemic lupus erythematosus (SLE) despite stable standard of care (SOC) medication defined as:

  a. Diagnosed with SLE at least 24 weeks before the Screening Visit (Visit 1) study entry by a qualified physician b. Classified by 2019 SLE European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE c. With serological evidence for SLE at Screening as demonstrated by at least 1 of the following: i) Evidence for anti-dsDNA (in central laboratory at Screening) ii) Either complement C3 < lower limit of normal (LLN) OR complement C4 <LLN OR elevated erythrocyte-bound complement C4d (where available) as measured by central laboratory iii) Antinuclear antibodies with a titer of at least 1:80 confirmed by central laboratory in combination with evidence of at least 1 of the following SLE typical autoantibodies:

  1. Anti-Smith (anti-Sm) antibodies (central laboratory) 2. Anti-Sjögren's syndrome antibody A (Anti-SSA) (Ro)/Anti-Sjögren's syndrome antibody B (anti-SSB) (La) autoantibodies (central laboratory) 3. Historic evidence for anti-dsDNA antibodies

  d. Moderately to severely active defined as
* British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) Grade B in ≥2 organ systems and/or a BILAG 2004 Grade A in ≥1 organ systems at Screening and Baseline Visit AND
* Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≥6 at Screening Visit AND
* SLEDAI-2K without labs ≥4 at Baseline Visit

  e. Receiving the following SOC medication at stable dose:
  * Antimalarial treatment in combination with corticosteroids and/or immunosuppressants or as stand-alone treatment if justified OR Treatment with corticosteroids and/or immunosuppressants if anti-malarial treatment is not possible

Exclusion Criteria:

* Study participant has any medical or psychiatric condition (including conditions due to neuropsychiatric systemic lupus erythematosus (SLE)) that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study. This includes study participants with a life threatening condition
* Study participant has a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins, or monoclonal antibodies
* Study participant has a history of malignancy, except the following treated cancers: cervical carcinoma in situ, basal cell carcinoma, or dermatological squamous cell carcinoma
* Study participant has an increased risk for thromboembolic events due to an ongoing heart disease or due to a medical device, including but not limited to vascular graft, valvular heart disease, atrial fibrillation, or a heart rhythm disorder
* Study participant has evidence of human immunodeficiency virus (HIV) infection, agammaglobulinemias, T-cell deficiencies, or human T-cell lymphotropic virus-1 infection
* Study participant had a reactivated latent infection (example, cytomegalovirus, herpes simplex virus, or herpes zoster infection) or opportunistic infection (including but not limited to, pneumocystis, cytomegalovirus, or severe herpes zoster infection) within 12 weeks prior to the first study medication infusion (Visit 2), or is currently receiving suppressive therapy for an opportunistic infection
* Study participants who have received live/live attenuated vaccines within 6 weeks prior to the first study medication infusion
* Study participant has clinically significant active or latent infection
* Study participant has a mixed connective tissue disease, scleroderma, and/or overlap syndrome of these diseases with SLE
* Study participant takes any protocol defined prohibited concomitant medication
* Study participant has previously been randomized within this study or participant has previously been assigned to treatment with dapirolizumab pegol (DZP) in a study evaluating DZP
* Study participant has participated in another study of an IMP within the previous 12 weeks or 5 half-lives of the investigational medicinal product (IMP) whatever is longer or is currently participating in another study of an IMP
* Study participant has chronic kidney failure stage 4, manifested by estimated glomerular filtration rate <30mL/min/1.73m^2, or serum creatinine >2.5 mg/dL, or participant has proteinuria >3 g/day, or protein: creatinine ratio >340 mg/mmol at the Screening Visit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (177):
- United States (60):
  - Sl0043 50140, Birmingham, Alabama
  - Sl0043 50052, Phoenix, Arizona
  - Sl0043 50328, Tucson, Arizona
  - Sl0043 50383, Beverly Hills, California
  - Sl0043 50257, La Jolla, California
  - Sl0043 50275, La Palma, California
  - Sl0043 50378, Loma Linda, California
  - Sl0043 50258, Los Angeles, California
  - Sl0043 50340, Orange, California
  - Sl0043 50331, Poway, California
  - Sl0043 50377, San Diego, California
  - Sl0043 50316, San Leandro, California
  - Sl0043 50339, Denver, Colorado
  - Sl0043 50367, New Haven, Connecticut
  - Sl0043 50341, Washington D.C., District of Columbia
  - Sl0043 50239, Brandon, Florida
  - Sl0043 50362, Gainesville, Florida
  - Sl0043 50122, Miami, Florida
  - Sl0043 50059, Ormond Beach, Florida
  - Sl0043 50324, Plantation, Florida
  - Sl0043 50329, Tampa, Florida
  - Sl0043 50283, Tampa, Florida
  - Sl0043 50368, Atlanta, Georgia
  - Sl0043 50382, Atlanta, Georgia
  - Sl0043 50240, Idaho Falls, Idaho
  - Sl0043 50310, Chicago, Illinois
  - Sl0043 50360, Skokie, Illinois
  - Sl0043 50474, Hopkinsville, Kentucky
  - Sl0043 50285, Lake Charles, Louisiana
  - Sl0043 50288, Cumberland, Maryland
  - Sl0043 50015, Hagerstown, Maryland
  - Sl0043 50219, Detroit, Michigan
  - Sl0043 50333, Grand Blanc, Michigan
  - Sl0043 50273, Las Vegas, Nevada
  - Sl0043 50010, Brooklyn, New York
  - Sl0043 50366, Canton, New York
  - Sl0043 50266, Great Neck, New York
  - Sl0043 50264, Manhasset, New York
  - Sl0043 50077, New York, New York
  - Sl0043 50334, New York, New York
  - Sl0043 50241, Syracuse, New York
  - Sl0043 50238, Charlotte, North Carolina
  - Sl0043 50179, Winston-Salem, North Carolina
  - Sl0043 50330, Cincinnati, Ohio
  - Sl0043 50262, Oklahoma City, Oklahoma
  - Sl0043 50020, Duncansville, Pennsylvania
  - Sl0043 50147, Hershey, Pennsylvania
  - Sl0043 50364, Philadelphia, Pennsylvania
  - Sl0043 50365, Pittsburgh, Pennsylvania
  - Sl0043 50001, Jackson, Tennessee
  - Sl0043 50263, Amarillo, Texas
  - Sl0043 50338, Bellaire, Texas
  - Sl0043 50418, Colleyville, Texas
  - Sl0043 50057, Dallas, Texas
  - Sl0043 50304, Dallas, Texas
  - Sl0043 50036, Mesquite, Texas
  - Sl0043 50267, Seattle, Washington
  - Sl0043 50061, Spokane, Washington
  - Sl0043 50050, Beckley, West Virginia
  - Sl0043 50321, Morgantown, West Virginia
- Argentina (7):
  - Sl0043 60002, Capital Federal
  - Sl0043 60001, Ciudad Autonoma de Buenos AIRE
  - Sl0043 60029, Mendoza
  - Sl0043 60003, Quilmes
  - Sl0043 60022, Quilmes
  - Sl0043 60011, San Juan
  - Sl0043 60014, San Miguel de Tucumán
- Australia (2):
  - Sl0043 30020, Parkville
  - Sl0043 30025, St Albans
- Austria (2):
  - Sl0043 40388, Graz
  - Sl0043 40387, Vienna
- Belgium (2):
  - Sl0043 40123, Brussels
  - Sl0043 40060, Liège
- Bulgaria (4):
  - Sl0043 40006, Plovdiv
  - Sl0043 40189, Plovdiv
  - Sl0043 40522, Plovdiv
  - Sl0043 40380, Sofia
- Canada (5):
  - Sl0043 50374, Calgary
  - Sl0043 50337, Edmonton
  - Sl0043 50259, Rimouski
  - Sl0043 50045, Toronto
  - Sl0043 50044, Trois-Rivières
- Chile (4):
  - Sl0043 60021, Providencia, Santiago
  - Sl0043 60015, Santiago
  - Sl0043 60018, Santiago
  - Sl0043 60030, Santiago
- Colombia (8):
  - Sl0043 60013, Barranquilla
  - Sl0043 60019, Barranquilla
  - Sl0043 60006, Bogotá
  - Sl0043 60027, Bogotá
  - Sl0043 60016, Bucaramanga
  - Sl0043 60007, Chía
  - Sl0043 60028, Medellín
  - Sl0043 60031, Montería
- Sl0043 40066, Prague, Czechia
- Sl0043 40489, Odense, Denmark
- France (2):
  - Sl0043 40506, Montpellier
  - Sl0043 40505, Paris
- Germany (8):
  - Sl0043 40386, Cologne
  - Sl0043 40322, Dessau
  - Sl0043 40356, Dresden
  - Sl0043 40072, Freiburg im Breisgau
  - Sl0043 40024, Hanover
  - Sl0043 40027, Herne
  - Sl0043 40078, Leipzig
  - Sl0043 40402, Tübingen
- Greece (5):
  - Sl0043 40378, Athens
  - Sl0043 40377, Crete
  - Sl0043 40501, Haidari - Athens
  - Sl0043 40507, Larissa
  - Sl0043 40375, Thessaloniki
- Hungary (5):
  - Sl0043 40412, Budapest
  - Sl0043 40411, Debrecen
  - Sl0043 40413, Gyula
  - Sl0043 40031, Szeged
  - Sl0043 40499, Székesfehérvár
- Italy (9):
  - Sl0043 40084, Catania
  - Sl0043 40472, Ferrara
  - Sl0043 40514, Genova
  - Sl0043 40291, Milan
  - Sl0043 40448, Milan
  - Sl0043 40471, Milan
  - Sl0043 40509, Padua
  - Sl0043 40148, Roma
  - Sl0043 40492, Rozzano
- Mexico (6):
  - Sl0043 50317, Chihuahua City
  - Sl0043 50250, Cuernavaca
  - Sl0043 50249, Guadalajara
  - Sl0043 50271, León
  - Sl0043 50252, Mérida
  - Sl0043 50251, Monterrey
- Peru (4):
  - Sl0043 60026, Arequipa
  - Sl0043 60008, Lima
  - Sl0043 60009, Lima
  - Sl0043 60023, Lima
- Philippines (4):
  - Sl0043 20110, Angeles
  - Sl0043 20182, Davao City
  - Sl0043 20181, Makati
  - Sl0043 20111, Manila
- Poland (15):
  - Sl0043 40482, Bialystok
  - Sl0043 40119, Bydgoszcz
  - Sl0043 40398, Katowice
  - Sl0043 40490, Krakow
  - Sl0043 40502, Krakow
  - Sl0043 40037, Lublin
  - Sl0043 40151, Lublin
  - Sl0043 40483, Nadarzyn
  - Sl0043 40044, Poznan
  - Sl0043 40090, Poznan
  - Sl0043 40097, Warsaw
  - Sl0043 40098, Warsaw
  - Sl0043 40394, Warsaw
  - Sl0043 40397, Wroclaw
  - Sl0043 40481, Wroclaw
- Romania (3):
  - Sl0043 40383, Bucharest
  - Sl0043 40464, Bucharest
  - Sl0043 40382, Galati
- Serbia (4):
  - Sl0043 40393, Belgrade
  - Sl0043 40461, Belgrade
  - Sl0043 40466, Kragujevac
  - Sl0043 40392, Novi Sad
- South Korea (4):
  - Sl0043 20141, Busan
  - Sl0043 20106, Daejeon
  - Sl0043 20108, Incheon
  - Sl0043 20104, Seoul
- Spain (7):
  - Sl0043 40045, A Coruña
  - Sl0043 40160, Barcelona
  - Sl0043 40341, Málaga
  - Sl0043 40521, Mérida
  - Sl0043 40101, Sabadell
  - Sl0043 40400, Seville
  - Sl0043 40099, Vigo
- Taiwan (5):
  - Sl0043 20113, Taichung
  - Sl0043 20142, Taichung
  - Sl0043 20095, Taipei
  - Sl0043 20099, Taipei
  - Sl0043 20082, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2020 and concluded in June 2024.
Pre-assignment Details: Participant flow refers to the Randomized Set (RS).
Groups:
- PBO+SOC: Participants received placebo (PBO) as an intravenous (iv) infusion every 4 weeks (Q4W) in combination with Standard of Care (SOC) during 48 weeks Treatment Period.
- DZP+SOC: Participants received Dapirolizumab pegol (DZP) 24 milligrams/kilogram (mg/kg) as an iv infusion Q4W in combination with SOC during 48 weeks Treatment Period.
Period: Overall Study
Arm/Group | PBO+SOC | DZP+SOC
Started | 108 | 213
Completed | 91 | 192
Not Completed | 17 | 21
Not completed — Lack of Efficacy | 4 | 4
Not completed — Consent Withdrawal by Study Participant | 9 | 7
Not completed — Patient has a Renal Flare | 1 | 0
Not completed — SLE Worsening | 0 | 1
Not completed — Subject Decision due to Personal Reason | 0 | 1
Not completed — PI closed Site - Subject Early Withdrawal | 0 | 1
Not completed — Subject Withdrew due to Personal Reason | 0 | 1
Not completed — Subject Moved to Another State | 0 | 1
Not completed — Adverse event, serious fatal | 0 | 1
Not completed — Adverse event, non-fatal | 3 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all study participants who were randomized and had received at least 1 dose (any amount) of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO+SOC | DZP+SOC | Total
Number analyzed (Participants) | 108 | 213 | 321
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.5 (12.3) | 43.8 (12.4) | 43.0 (12.4)
Age, Customized [Count of Participants; unit: Participants]
  12 to <18 Years | 0 | 1 | 1
  18 to <65 Years | 106 | 201 | 307
  65 to <85 Years | 2 | 11 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 198 | 299
  Male | 7 | 15 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska native | 9 | 20 | 29
  Asian | 9 | 18 | 27
  Black or African American | 10 | 14 | 24
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White | 63 | 130 | 193
  Other/Mixed | 17 | 30 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 78 | 118
  Not Hispanic or Latino | 68 | 135 | 203

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Achievement of BILAG 2004-based Composite Lupus Assessment (BICLA) Response at Week 48
Description: Study participants were considered to be a BILAG 2004-based Composite Lupus Assessment (BICLA) responder if all of the following were fulfilled:
  * British Isles Lupus Assessment Group Disease Activity Index 2004 (BILAG 2004) improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and less than or equal to [≤] 1 new B.); Here, score A ("Active"): Severely active disease; score B ("Beware"): Moderately active disease; score C ("Contentment"): Mild stable disease; score D ("Discount"): Inactive now but previously active; and
  * No worsening in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  * No worsening in the Physician's Global Assessment of Disease (PGA) compared to Baseline Visit defined as [≤] 10 millimeter (mm) increase on a 100 mm visual analog scale (VAS).
Time Frame: Week 48
Population: The Full Analysis Set (FAS) consisted of all study participants randomized into the study except 6 participants excluded from FAS due to persistent Good Clinical Practice (GCP) non-compliance at the site enrolling them.
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 34.6 | 49.5
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority — The difference in proportion responding between SOC+DZP 24mg/kg and SOC+PBO was estimated and tested using the Cochran-Mantel-Haenszel (CMH) risk difference estimate controlling for the randomization stratification factors, Pooled Region (North America vs Western Europe/Asia-Pacific vs Latin America/Eastern Europe), Screening disease activity (chronic active vs acute flaring) and Screening SLEDAI score (<10 vs >=10); p = 0.0110, Cochran-Mantel-Haenszel; Difference in Proportions (%) = 14.6, 95% CI 2-sided [3.3 to 25.8]

2. Secondary Outcome: Percentage of Participants With Achievement of BICLA Response at Week 24
Description: Study participants were considered to be a BICLA responder if all of the following were fulfilled:
  * BILAG 2004 improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤ 1 new B.); Here, score A ("Active"): Severely active disease; score B ("Beware"): Moderately active disease; score C ("Contentment"): Mild stable disease; score D ("Discount"): Inactive now but previously active; and
  * No worsening in the SLEDAI-2K total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  * No worsening in the PGA compared to Baseline Visit defined as ≤ 10 mm increase on a 100 mm VAS.
Time Frame: Week 24
Population: The FAS consisted of all study participants randomized into the study except 6 participants excluded from FAS due to persistent GCP non-compliance at the site enrolling them.
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 38.3 | 46.6
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority — The difference in proportion responding between SOC+DZP 24mg/kg and SOC+PBO was estimated and tested using the CMH risk difference estimate controlling for the randomization stratification factors, Pooled Region (North America vs Western Europe/Asia-Pacific vs Latin America/Eastern Europe), Screening disease activity (chronic active vs acute flaring) and Screening SLEDAI score (<10 vs >=10); p = 0.1776, Cochran-Mantel-Haenszel; Difference in Proportions (%) = 7.9, 95% CI 2-sided [-3.6 to 19.4]

3. Secondary Outcome: Percentage of Participants With Achievement of BICLA Response at Week 12
Description: Study participants were considered to be a BICLA responder if all of the following were fulfilled:
  * BILAG 2004 improvement without worsening (A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤ 1 new B.); Here, score A ("Active"): Severely active disease; score B ("Beware"): Moderately active disease; score C ("Contentment"): Mild stable disease; score D ("Discount"): Inactive now but previously active and
  * No worsening in the SLEDAI-2K total score compared to Baseline Visit (defined as no increase in SLEDAI-2K total score); and
  * No worsening in the PGA compared to Baseline Visit defined as ≤ 10 mm increase on a 100 mm VAS.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 29.0 | 39.9
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0518, Cochran-Mantel-Haenszel; Difference in Proportions (%) = 10.8, 95% CI 2-sided [-0.1 to 21.7]

4. Secondary Outcome: Percentage of Participants With Achievement of Prevention of Severe British Isles Lupus Assessment Group (BILAG) Flares (Severe BILAG Flare-free) Through Week 48
Description: A severe BILAG flare was defined as a british isles lupus assessment group disease activity index 2004 (BILAG 2004) Grade A in any system due to individual items that were new or worse qualifying for the Grade A. Determination of items that were new or worse and were qualifying for the Grade A were according to the supplementary information for the numerical scoring of the BILAG-2004 index. Here, Grade A ("Active"): Severely active disease (sufficient to require systemic immunosuppressant or anticoagulant therapy.
Time Frame: During Treatment Period up to Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 76.6 | 88.4
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0257, Cochran-Mantel-Haenszel; Difference in Proportions (%) = 11.5, 95% CI 2-sided [1.4 to 21.6]

5. Secondary Outcome: Percentage of Participants With Achievement of Lupus Low Disease Activity State (LLDAS) in ≥50% of Post-Baseline Visits Through Week 48
Description: The LLDAS includes domains that capture the absence of organ-threatening disease activity and harmful treatment burden. The LLDAS is defined as:
  * SLEDAI-2K score was ≤4 with no activity in major organ systems.
  * No new and/or worsening disease activity defined as no SLEDAI-2K component documented as present that was not documented present at the previous visit.
  * PGA ≤ 33 mm.
  * Prednisone equivalent systemic dose for systemic lupus erythematosus (SLE) indication ≤ 7.5 mg per day.
  * Stable standard maintenance doses of immunosuppressive drugs as allowed by protocol, defined as no increase in dose in the past 12 weeks and no dose higher than allowed as per protocol.
Time Frame: During Treatment Period up to Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 15.9 | 23.6
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1042, Cochran-Mantel-Haenszel; Difference in Proportions (%) = 7.2, 95% CI 2-sided [-1.5 to 16.0]

6. Secondary Outcome: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) at Week 48
Description: The SLEDAI-2K is a global index which includes 24 clinical and laboratory variables such as antibodies, renal, and hematological components measured 30 days before, and at the timepoint of assessment. The variables were weighted by the type of manifestation, but not by severity or dynamic of the individual item. The SLEDAI-2K includes scoring for antibodies (anti-dsDNA positive or negative) and low complement, as well as some renal and hematologic parameters. The total score falls between 0 and 105, with higher scores representing increased disease activity. Mixed effects models for repeated measurements (MMRM).
Time Frame: From Baseline (Day 1) to Week 48
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
score on a scale | -4.2 (0.39) | -6.1 (0.26)
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority; p = 0.0001, MMRM; The Least Squares (LS) Mean, the difference (DZP+SOC versus PBO+SOC), and the 95% CIs was computed from the MMRM; Difference of Change(DZP+SOC vs PBO+SOC) = -1.8, 95% CI 2-sided [-2.7 to -0.9]

7. Secondary Outcome: Percentage of Participants With Achievement of BILAG Improvement Without Worsening at Week 48
Description: The BILAG improvement without worsening defined as A scores at Baseline improved to B, C or D; B scores improved to C or D; no new A scores and ≤1 new B Score. Here, score A ("Active"): Severely active disease (sufficient to require systemic immunosuppressant or anticoagulant therapy; score B ("Beware"): Moderately active disease (requires low dose or local immunosuppressant therapy or symptomatic therapy; score C ("Contentment"): Mild stable disease (no indication for changes in treatment); score D ("Discount"): Inactive now but previously active.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 34.6 | 49.5

8. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PGA) at Week 48
Description: The PGA is a measure of systemic lupus erythematosus (SLE) signs and symptoms by the physician using a visual analog scale of 0 to 100mm, Where 0 indicate "very good", asymptomatic, and no limitation of normal activity and 100 indicate "severe disease".
Time Frame: From Baseline (Day 1) to Week 48
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
score on a scale | -33.4 (1.99) | -39.6 (1.36)

9. Secondary Outcome: Percentage of Participants With Achievement of Systemic Lupus Erythematosus Responder Index Response - 4 (SRI-4) Response at Week 48
Description: The SRI-4 define responders as meeting all of the following criteria:
  * Reduction in SLEDAI-2K score of ≥ 4.
  * No shift from BILAG 2004 Grade B, C, D, or E to A post-Baseline. Here, Grade A ("Active"): Severely active disease; Grade B ("Beware"): Moderately active disease; Grade C ("Contentment"): Mild stable disease; Grade D ("Discount"): Inactive now but previously active; Grade E ("Excluded"): Never affected.
  * No more than 1 shift from BILAG 2004 Grade C, D, or E to B post-Baseline.
  * No worsening in the PGA compared to study entry defined as ≤ 10 mm increase on a 100 mm visual analog scale, equivalent to less than a 10 mm increase in the PGA compared to study entry score.
Time Frame: Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 41.1 | 60.1

10. Secondary Outcome: Percentage of Participants With Achievement of Prevention of Moderate/Severe BILAG Flares (Moderate/Severe BILAG Flare-free) Through Week 48
Description: Achievement of prevention of moderate/severe BILAG flares through Week 48 was defined as the percentage of participants with no moderate or severe flare through Week 48. A severe BILAG flare was defined as a BILAG 2004 Grade A in any system due to individual items that were new or worse qualifying for the Grade A. Determination of items that were new or worse and were qualifying for the Grade A, according to the supplementary information for the numerical scoring of the BILAG-2004 index. A moderate BILAG flare was defined as 2 or more BILAG 2004 Grade B due to individual items that were new or worse and were qualifying for the Grade B in any system. Determination of items that were new or worse qualifying for the Grade B, according to the supplementary information for the numerical scoring of the BILAG- 2004 index. Here, Grade A ("Active"): Severely active disease; Grade B ("Beware"): Moderately active disease.
Time Frame: During Treatment Period up to Week 48
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
percentage of participants | 63.0 | 78.6

11. Secondary Outcome: Time to Severe BILAG Flare Through Week 48
Description: Time to severe BILAG flare (the event) through Week 48 was defined as the time from randomization until the start of the event. A severe BILAG flare was defined as a BILAG 2004 Grade A in any system due to individual items that were new or worse qualifying for the Grade A. Determination of items that were new or worse and were qualifying for the Grade A, according to the supplementary information for the numerical scoring of the BILAG-2004 index. Here, Grade A ("Active"): Severely active disease.
Time Frame: During Treatment Period up to Week 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
weeks | NA [NA to NA] — The time to flare estimate of the 25 percentile, median, 75 percentile time could not be calculated and presented due to the low number of events (less than 25%, 50%, 75% participants respectively had flare events in this arm). | NA [NA to NA] — The time to flare estimate of the 25 percentile, median, 75 percentile time could not be calculated and presented due to the low number of events (less than 25%, 50%, 75% participants respectively had flare events in this arm).
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority; p = 0.0111, Log Rank

12. Secondary Outcome: Time to Moderate/Severe BILAG Flare Through Week 48
Description: Time to moderate/severe BILAG flare (the event) through Week 48 was defined as the time from randomization until the start of the event. Moderate BILAG flare was defined as 2 or more BILAG 2004 Grade B due to individual items that were new or worse and were qualifying for the Grade B in any system. Determination of items that were new or worse qualifying for the Grade B, according to the supplementary information for the numerical scoring of the BILAG-2004 index. Severe BILAG flare was defined as a BILAG 2004 Grade A in any system due to individual items that were new or worse qualifying for the Grade A. Determination of items that were new or worse and are qualifying for the Grade A, according to the supplementary information for the numerical scoring of the BILAG-2004 index. Here, Grade A ("Active"): Severely active disease; Grade B ("Beware"): Moderately active disease.
Time Frame: During Treatment Period up to Week 48
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 107 | 208
weeks | NA [36.1 to NA] — The time to flare estimate of the median, 75 percentile time could not be calculated and presented due to the low number of events (less than 50% and 75% participants respectively had flare events in this arm). | NA [NA to NA] — The time to flare estimate of the 25 percentile, median, 75 percentile time could not be calculated and presented due to the low number of events (less than 25%, 50%, 75% participants respectively had flare events in this arm).
Statistical Analysis 1: Comparison: PBO+SOC vs DZP+SOC; Test type: Superiority; p = 0.0228, Log Rank

13. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP. Treatment-emergent AEs were those with onset date on or after the first administration of study drug, and up to 60 days after last dose.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 54)
Population: The SS consisted of all study participants who were randomized and had received at least 1 dose (any amount) of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 108 | 213
percentage of participants | 75.0 | 82.6

14. Secondary Outcome: Percentage of Participants With Serious Treatment-emergent Adverse Events During the Study
Description: A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: Results in death; Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization; Results in persistent disability/incapacity; Is a congenital anomaly/birth defect; and Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above. Treatment-emergent AEs were those with onset date on or after the first administration of study drug, and up to 60 days after last dose.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 54)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 108 | 213
percentage of participants | 14.8 | 9.9

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Special Interest During the Study
Description: An adverse event of special interest (AESIs) is any AE that a regulatory authority has mandated be reported on an expedited basis, regardless of the seriousness, expectedness, or relatedness of the AE to the administration of a product/compound.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 54)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 108 | 213
percentage of participants | 0.9 | 0

16. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Special Monitoring During the Study
Description: An AE of special monitoring is a product-specific AEs, adverse reactions, or safety topics considered as requiring special monitoring by UCB.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 54)
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | PBO+SOC | DZP+SOC
Number analyzed (Participants) | 108 | 213
percentage of participants | 24.1 | 36.6

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 54)
Description: Treatment-emergent AEs were those with onset date on or after the first administration of study drug, and up to 60 days after last dose. The SS consisted of all study participants who were randomized and had received at least 1 dose (any amount) of study medication.
Arm/Group | PBO+SOC | DZP+SOC
All-Cause Mortality (participants affected / at risk) | 0/108 | 1/213
Serious Adverse Events (participants affected / at risk) | 16/108 | 21/213
Other Adverse Events (participants affected / at risk) | 47/108 | 109/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO+SOC (N=108) | DZP+SOC (N=213)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Lupus myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lupus enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 2 (2) — The two events were reported as "herpes zoster over left eyelid and forehead, V1" and "left herpes zoster ophthlamicus (dermatome V1/V2).
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Joint tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — The AE of suicidal ideation occurred before administration of the first dose of study treatment. Only for technical reasons it was listed in the analysis as "treatment emergent" as the onset date was the day of first study treatment.
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shrinking lung syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBO+SOC (N=108) | DZP+SOC (N=213)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 15 (15)
Nausea (Gastrointestinal disorders) | 6 (9) | 9 (9)
COVID-19 (Infections and infestations) | 17 (18) | 44 (44)
Herpes zoster (Infections and infestations) | 6 (7) | 4 (4)
Oral herpes (Infections and infestations) | 6 (8) | 4 (4)
Bronchitis (Infections and infestations) | 5 (6) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 20 (23)
Nasopharyngitis (Infections and infestations) | 13 (19) | 18 (23)
Urinary tract infection (Infections and infestations) | 9 (10) | 28 (36)
Headache (Nervous system disorders) | 7 (8) | 15 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04294667/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04294667/SAP_001.pdf